CLINICAL TRIAL: NCT04174560
Title: Phase I Study to Determine the Optimal Human Challenge Dose for Norovirus GII.4 CIN-3 Batch No.: 01-16C3
Brief Title: Phase I Norovirus Challenge Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: 17-0102
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-01-03

CONDITIONS: Gastroenteritis Norovirus
Keywords: Healthy Adults; Norovirus GII.4 CIN-3; Optimal Human Challenge Dose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Single dose (3.5x10^3 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given orally to subjects with functional FUT-2 gene (secretor positive), n=15, and single dose (3.5x10^3 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given to subjects with a lack a non-functional FUT-2 gene (non-secretor), n=1, on Day 1
  Interventions: Biological: Norovirus GII.4 Challenge Pool
- Cohort 2 (Experimental): Single dose (3.5x10^4 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given orally to subjects with functional FUT-2 gene (secretor positive), n=15, and single dose (3.5x10^4 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given to subjects with a lack a non-functional FUT-2 gene (non-secretor), n=1, on Day 1
  Interventions: Biological: Norovirus GII.4 Challenge Pool
- Cohort 3 (Experimental): Single dose (3.5x10^5 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given orally to subjects with functional FUT-2 gene (secretor positive), n=15, and single dose (3.5x10^5 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given to subjects with a lack a non-functional FUT-2 gene (non-secretor), n=1, on Day 1
  Interventions: Biological: Norovirus GII.4 Challenge Pool

INTERVENTIONS:
Biological: Norovirus GII.4 Challenge Pool — Subjects will be NPO (nothing by mouth) for at least 90 minutes followed by ingestion of 60 mL of a 2% sodium bicarbonate solution by mouth. 2 minutes later, subjects will be administered Norovirus GII.4 CIN-3. Five minutes following administration of the challenge dose, subjects will be administered a 60 mL volume of a 2% sodium bicarbonate solution and then remain NPO for at least the next 90 minutes. Subjects will be observed during the 60 minutes after receipt of the challenge by a study team member to detect and treat any immediate adverse reactions.

SUMMARY:
This is a safety and infectivity study of experimental human Norovirus genogroup GII.4 administered to 48 healthy non-pregnant adults, 18-49 years of age, negative for COVID-19 by antigen testing at the time of norovirus challenge. Subjects will be admitted to the Vaccine Research Center inpatient facility and challenged with a dose of human norovirus GII.4 challenge strain. The challenge study will be conducted in 3 cohorts of approximately 16 subjects each, 15 subjects will have a functional FUT-2 gene (secretor positive) and 1 subject will have a non-functional FUT-2 gene (non-secretor). Subjects in Cohort 1 will receive 3.5x10^3 copies of norovirus, in Cohort 2 will receive 3.5x10^4 copies of norovirus and in Cohort 3 will receive 3.5x10^5 copies of norovirus. Based on the illness rate of subjects meeting the primary outcome measure in secretor - positive subjects of the initial cohort, the decision will be made with regards to dosing of the second and the third cohorts. Study duration is approximately 12-18 months with subject participation duration of 6-8 months. The primary objective of this study is to determine the optimal challenge dose of Norovirus GII.4 CIN-3 Batch No.: 01-16C3 to achieve illness in > / = 50% of subjects (illness is defined as norovirus infection determined by positive Polymerase Chain Reaction (PCR) and either: a) > / = 3 loose or liquid stools, in a 24-hour period, b) > / = 300 gm of loose or liquid stool in a 24-hour period or c) and/or any episode of vomiting), during the inpatient period.

DETAILED DESCRIPTION:
This is a double-blind, safety and infectivity study of experimental human Norovirus genogroup GII.4 administered to 48 healthy non-pregnant adults, 18-49 years of age, negative for COVID-19 by antigen testing at the time of norovirus challenge. Subjects will be admitted to the Vaccine Research Center inpatient facility and challenged with a dose of human norovirus GII.4 challenge strain. The challenge study will be conducted in 3 cohorts of approximately 16 subjects each, 15 subjects will have a functional FUT-2 gene (secretor positive) and 1 subject will have a non-functional FUT-2 gene (non-secretor). Subjects in Cohort 1 will receive 3.5x10^3 copies of norovirus, in Cohort 2 will receive 3.5x10^4 copies of norovirus and in Cohort 3 will receive 3.5x10^5 copies of norovirus. Based on the illness rate of subjects meeting the primary outcome measure in secretor - positive subjects of the initial cohort, the decision will be made with regards to dosing of the second and the third cohorts. Subjects will remain in the inpatient facility for at least four days following the challenge and assessed daily for clinical and virologic evidence of norovirus infection. After the discharge, subjects will return to the site for evaluation on Days 6, 15, 30, 45, and 60 post challenge. A final phone call will be performed at day 180 to obtain an interim medical history. Study duration is approximately 12-18 months with subject participation duration of 6-8 months. The primary objective of this study is to determine the optimal challenge dose of Norovirus GII.4 CIN-3 Batch No.: 01-16C3 to achieve illness in > / = 50% of subjects (illness is defined as norovirus infection determined by positive Polymerase Chain Reaction (PCR) and either: a) > / = 3 loose or liquid stools, in a 24-hour period, b) > / = 300 gm of loose or liquid stool in a 24-hour period or c) and/or any episode of vomiting), during the inpatient period. The secondary objectives are: 1) To evaluate the safety of the Norovirus GII.4 CIN-3 Batch No.: 01-16C3 challenge strain; 2) To determine the rate of infection at different challenge doses by detection of norovirus GII.4 in the stool using specific qRT-PCR and Anti-norovirus GII.4 serum IgG by Enzyme-Linked Immunnosorbent Assay (ELISA) (> / = 4-fold rise from baseline through Day 30); 3) To measure the severity of acute gastroenteritis; 4) To determine the quantity and duration of virus shedding in stool by qRT-PCR.

ELIGIBILITY:
Inclusion Criteria:

1. Subject able to provide informed consent.
2. Male or non-pregnant females between the ages of 18 and 49 years, inclusive.
3. Women of childbearing potential must be using an acceptable method of birth control for at least 30 days prior to enrollment through day 45 after receipt of challenge virus.

   * A woman is considered of childbearing potential unless post-menopausal (absence of menses for > / = 1 year) or surgically sterilized (tubal ligation, bilateral oophorectomy or hysterectomy).
   * Acceptable contraception methods for women include but are not limited to: sexual abstinence from intercourse with men, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject enrolling in the study, barrier methods such as condoms or diaphragms with spermicide or foam, effective devices (intrauterine devices (IUD's), NuvaRing (R)) or licensed hormonal products such as implants, injectables or oral contraceptives.
4. For women of childbearing potential, must have a negative serum or urine pregnancy test at screening.
5. Are in good general health*.

   *As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, Emergency Room (ER), or urgent care for condition and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination.
6. Demonstrate knowledge and comprehension of the study by scoring > / = 70% on a quiz (test of understanding) of the study protocol and policies.
7. Willing and able to participate in all study visits, including an inpatient stay of at least 96 hours.

Exclusion Criteria:

1. Have household contact with or have daily contact with children less than 2 years of age or persons older than 70 years of age.
2. Have expected extended social contact (> 2 hours/day) with immunocompromised individuals in the 8 weeks after challenge*.

   *Including persons with HIV infection or active cancer, children <2 years of age, pregnant women or persons who are immunosuppressed (e.g. history of stem cell or organ transplantation) and/or provide any child day care services (in-home or non-residential facility).
3. Are healthcare workers with direct patient contact or any child day care services (in-home or non-residential facility) in the 8 weeks after challenge.
4. Are positive for COVID-19 by an antigen test at the time of admission to the challenge unit.
5. Are food service workers expected to prepare/handle food in the 8 weeks after challenge.
6. Plan to be living in a confined communal environment (e.g. ship, camp, or dormitory) within 8 weeks after receiving the challenge strain.
7. For females, are pregnant or plan to become pregnant at any time between the Screening Visit through 45 days after receipt of the challenge virus.
8. Are breastfeeding or plan to breastfeed at any given time throughout the study.
9. Have a history of acute gastroenteritis in the 4 weeks prior to challenge or any history of chronic or recurrent diarrhea or vomiting.
10. History of significant GI condition. *

    *Including: malabsorption, major GI surgery, current *eating disorder, irritable bowel syndrome, or any GI disorder (deemed clinically significant by study physician) making it unsafe to participate.
11. Have significant acute illness or an oral temperature > /= 100.4 degrees Fahrenheit within seven days prior to challenge.
12. Have a heart rate <45 beats per minute (bpm) or >100 bpm*.

    *If heart rate is <45 beats per minute and the investigator determines that this is not clinically significant (e.g., athletes) and heart rate increases > 45 beats per minute on moderate exercise (two flights of stairs), subject will not be excluded. If a subject has significant abnormalities in their heart rate, they will be informed of the values and advised to seek care from their physician.
13. Systolic blood pressure less than 90 mm Hg or greater than 150 mm Hg on two separate measurements (screening and baseline prior to challenge)*.

    *If a subject has significant abnormalities in their blood pressure, they will be informed of the values and advised to seek care from their physician.
14. Diastolic blood pressure less than 50 mm Hg or greater than 90 mm Hg on two separate measurements (screening and baseline, prior to challenge).
15. Have long-term use (> / = 2 weeks) of high-dose oral (> / = 20 mg per day prednisone or equivalent) or parenteral glucocorticoids, or high-dose inhaled steroids for greater than 7 days in the last 6 months.
16. Have an autoimmune, inflammatory, vasculitic or rheumatic disease, including but not limited to systemic lupus erythematosus, polymyalgia rheumatica, rheumatoid arthritis or scleroderma.
17. Have HIV, Hepatitis B, or Hepatitis C*.

    *Subjects will be tested for HIV, Hepatitis B surface antigen, and antibody to Hepatitis C at screening only. Any subjects having HIV, Hepatitis B, Hepatitis C infection will not be enrolled into the study.
18. Have a seizure disorder.
19. Have an active malignancy or history of malignancy* or current use of immunosuppressive or cytotoxic therapy.

    *Excluding nonmelanotic skin cancer in remission without treatment for more than 5 years.
20. Have abnormal screening laboratory test results per laboratory reported normal values*.

    *For white blood cells (WBCs), hemoglobin (Hgb), platelets, absolute neutrophil count (ANC), total bilirubin, potassium, sodium, and urine protein.
21. Serum creatinine greater than a Grade 1 adverse event on enrollment.
22. Alanine aminotransferase (ALT), greater than Grade 1 adverse event on enrollment.
23. Have a chronic condition that the study physician feels would pose a threat to participating subjects*.

    *Including, but not limited to solid organ or stem cell transplantation, diabetes, clinically significant history of immunosuppressive illness, gall bladder disease, heart disease, lung disease, pancreatic disease, renal disease or neurological disease.
24. Have ongoing drug abuse/dependence (including alcohol), or a history of these issues within 5 years of enrollment.
25. Have a positive urine test for opiates.
26. Have any medical, psychiatric, occupational, or behavioral problems that make it unlikely for the subject to comply with the protocol as determined by the investigator.
27. Are unwilling to comply with study procedures including abstaining from smoking for the duration of the inpatient portion of the study.
28. Have participated in a previous norovirus (NoV) challenge study or NoV vaccine study.
29. Have received experimental products within 30 days before study entry or plan to receive experimental products at any time during the study.
30. Plans to enroll in another clinical trial that could interfere with safety assessment of the investigational product at any time during the study period*.

    *Including study interventions such as drugs, biologics or devices.
31. Plan to donate blood during the course of the study.
32. Have received a live vaccine within 30 days before study entry or plan to receive a live vaccine prior to Day 30 of the study.
33. Have received, or plan to receive, an inactivated vaccine within 14 days of challenge to 14 days after challenge.
34. Received parenteral immunoglobulin or blood products within 3 months of challenge, or plan to receive parenteral immunoglobulin/blood products within 3 months after challenge.
35. Use of antibiotics within 7 days prior to entry into the inpatient facility.
36. Use of prescription and OTC medications containing acetaminophen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs within 48 hours prior to NoV challenge.
37. Regular use of laxatives or anti-motility agents.
38. Have a history of allergy to sodium bicarbonate.
39. Have had a recent norovirus infection or have ever had a norovirus vaccine.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy non-pregnant adults, 18-49 years of age, inclusive. They were recruited from the community at large around the clinical site. Participants were enrolled between 28MAR2022 and 10JUL2023.
Groups:
- 3.5x10^3 Copies - Secretor Positive: Single dose (3.5x10^3 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given orally to subjects with functional FUT-2 gene (secretor positive), on Day 1
  Norovirus GII.4 Challenge Pool: Subjects will be NPO (nothing by mouth) for at least 90 minutes followed by ingestion of 60 mL of a 2% sodium bicarbonate solution by mouth. 2 minutes later, subjects will be administered Norovirus GII.4 CIN-3. Five minutes following administration of the challenge dose, subjects will be administered a 60 mL volume of a 2% sodium bicarbonate solution and then remain NPO for at least the next 90 minutes. Subjects will be observed during the 60 minutes after receipt of the challenge by a study team member to detect and treat any immediate adverse reactions.
- 3.5x10^4 Copies - Secretor Positive: Single dose (3.5x10^4 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given orally to subjects with functional FUT-2 gene (secretor positive) on Day 1
  Norovirus GII.4 Challenge Pool: Subjects will be NPO (nothing by mouth) for at least 90 minutes followed by ingestion of 60 mL of a 2% sodium bicarbonate solution by mouth. 2 minutes later, subjects will be administered Norovirus GII.4 CIN-3. Five minutes following administration of the challenge dose, subjects will be administered a 60 mL volume of a 2% sodium bicarbonate solution and then remain NPO for at least the next 90 minutes. Subjects will be observed during the 60 minutes after receipt of the challenge by a study team member to detect and treat any immediate adverse reactions.
- 3.5x10^5 Copies - Secretor Positive: Single dose (3.5x10^5 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) will be given orally to subjects with functional FUT-2 gene (secretor positive), on Day 1
  Norovirus GII.4 Challenge Pool: Subjects will be NPO (nothing by mouth) for at least 90 minutes followed by ingestion of 60 mL of a 2% sodium bicarbonate solution by mouth. 2 minutes later, subjects will be administered Norovirus GII.4 CIN-3. Five minutes following administration of the challenge dose, subjects will be administered a 60 mL volume of a 2% sodium bicarbonate solution and then remain NPO for at least the next 90 minutes. Subjects will be observed during the 60 minutes after receipt of the challenge by a study team member to detect and treat any immediate adverse reactions.
- Secretor Negative: Single dose (3.5x10^3, 3.5x10^4 or 3.5x10^5 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) given orally. Participants lacked the secretor gene.
  Norovirus GII.4 Challenge Pool: Subjects will be NPO (nothing by mouth) for at least 90 minutes followed by ingestion of 60 mL of a 2% sodium bicarbonate solution by mouth. 2 minutes later, subjects will be administered Norovirus GII.4 CIN-3. Five minutes following administration of the challenge dose, subjects will be administered a 60 mL volume of a 2% sodium bicarbonate solution and then remain NPO for at least the next 90 minutes. Subjects will be observed during the 60 minutes after receipt of the challenge by a study team member to detect and treat any immediate adverse reactions.
Period: Overall Study
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Started | 15 | 12 | 18 | 3
Completed | 14 | 12 | 16 | 3
Not Completed | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3.5x10^3 Copies - Secretor Positive: Single dose (3.5x10^3 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) given orally. Participants tested positive for the secretor gene.
- 3.5x10^4 Copies - Secretor Positive: Single dose (3.5x10^4 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) given orally. Participants tested positive for the secretor gene.
- 3.5x10^5 Copies - Secretor Positive: Single dose (3.5x10^5 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) given orally. Participants tested positive for the secretor gene.
- Secretor Negative: Single dose (3.5x10^3, 3.5x10^4 or 3.5x10^5 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) given orally. Participants lacked the secretor gene.
- Total: Total of all reporting groups
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative | Total
Number analyzed (Participants) | 15 | 12 | 18 | 3 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (8.4) | 35.2 (7.7) | 35.3 (8.3) | 36.7 (8.5) | 36.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 14 | 1 | 26
  Male | 10 | 6 | 4 | 2 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 13 | 11 | 18 | 3 | 45
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 0 | 3 | 15
  White | 9 | 5 | 18 | 0 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 18 | 3 | 48

OUTCOME MEASURES:

1. Primary Outcome: The Occurrence of Norovirus-associated Illness in Secretor Positive Participants Through Day 4 After Challenge.
Description: Illness is defined as norovirus infection, determined by a positive PCR, and either a) = 3 loose or liquid stools in a 24-hour period, b) = 300 gm of loose or liquid stool in a 24-hour period, and/or c) any episode of vomiting.
Time Frame: Day 1 through Day 4
Population: Modified Intention-to-Treat Population: The mITT population includes all participants who received the challenge study product and contributed both pre- and at least one post-challenge sample during the inpatient period for which a conclusion can be made regarding illness and infectivity.
Measure: Count of Participants; unit: Participants
Groups:
- 3.5x10^3 Copies - Secretor Positive: Single dose (3.5x10^3 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) given orally
- 3.5x10^4 Copies - Secretor Positive: Single dose (3.5x10^4 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) given orally
- 3.5x10^5 Copies - Secretor Positive: Single dose (3.5x10^5 copies) of norovirus GII.4 CIN-3 Batch No.: 01-16C3 inoculum (with 60 mL of a 2% sodium bicarbonate before and after inoculum administration) given orally
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 15 | 12 | 18 | 3
Participants | 3 | 2 | 7 | 0

2. Secondary Outcome: The Number of Participants With Solicited Adverse Events Through Day 10
Description: Systemic solicited adverse events were collected pre-challenge, post-challenge, and via memory aid through 5 days after discharge from the isolation facility and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include headache, nausea, abdominal cramps/discomfort/pain, abdominal gurgling, abdominal bloating, myalgia, malaise/fatigue, anorexia/loss of appetite, and chills.
Time Frame: Day 1 through Day 10
Population: Safety Population: The Safety Analysis population includes all participants who received at least a partial dose of the challenge study product.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 15 | 12 | 18 | 3
Participants | 10 | 10 | 15 | 3

3. Secondary Outcome: The Number of Participants With Unsolicited Serious Adverse Events Reported Through Day 180.
Description: An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization (excluding any extended stay during challenge admission due to continued vomiting, diarrhea, etc.), a persistent or significant incapacity of substantial disruption of the ability to conduct normal life functions, a congenital anomaly/birth defect, important medical events that may not result in death, be life-threatening, or require hospitalizations may be considered serious when, based upon appropriate medical judgment they may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Day 180
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 15 | 12 | 18 | 3
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: The Number of Participants With Unsolicited Grade 3 Adverse Events From Challenge to Day 30
Description: ICH E6 defines an AE as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product. The FDA defines an AE as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Time Frame: Day 1 through Day 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 15 | 12 | 18 | 3
Participants | 0 | 0 | 2 | 0

5. Secondary Outcome: The Number of Participants With Infection Through Day 30
Description: Detection of norovirus GII.4 in stool by qRT-PCR at Days 2, 3, 4, 5, 6, 15, or 30; or >/= 4-fold rise from baseline in GII.4-specific antibody titers in serum IgG by ELISA through Day 30
Time Frame: Day 1 through Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 15 | 12 | 18 | 3
Participants
  Detection of norovirus GII.4 in stool | 4 | 4 | 9 | 0
  >/= 4-fold rise in GII.4-specific antibody titers in serum IgG | 3 | 4 | 9 | 1
  Norovirus GII.4 in stool OR >/= 4-fold rise in GII.4-specific antibody titers in serum IgG | 4 | 5 | 10 | 1

6. Secondary Outcome: Peak Genome Equivalent Copies/mL of Virus in Stool as Measured by qRT-PCR After Challenge Through Day 60
Description: Peak virus in stool as measured by qRT-PCR [genome equivalent copies per gram of stool (GEC/g)] is the maximum GEC/g of all available stool samples tested post-challenge.
Time Frame: Day 1 through Day 60
Population: Modified Intention-to-Treat Population: The mITT population includes all participants who received the challenge study product and contributed both pre- and at least one post-challenge sample during the inpatient period for which a conclusion can be made regarding illness and infectivity, restricted to participants who were shedding on at least one day.
Measure: Geometric Mean (95% Confidence Interval); unit: GEC/g
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 4 | 4 | 9 | 0
GEC/g | 230475280.31 [157130.618 to 338055406332] | 43569331.414 [156752.339 to 12110100882] | 176337339.33 [22259257.651 to 1396940442.9] |

7. Secondary Outcome: Duration (Number of Days) of Viral Secretion as Measured by qRT-PCR After Challenge Through Day 60
Description: Duration is based on the first and last days where norovirus is detected.
Time Frame: Day 1 through Day 60
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 4 | 4 | 9 | 0
Days | 5 (2.7) | 9.8 (11.7) | 3.9 (1.5) |

8. Secondary Outcome: Modified Vesikari Score Through Day 4
Description: The score is made up of the following components: duration of diarrhea (days), maximum number of diarrheal stools per 24 hours, duration of vomiting (days), maximum number of vomiting episodes per 24 hours, fever, and dehydration. Each of the components will be assigned a point value and the points will be summed to create a total score out of a possible 17 for each participant, with 17 being the worst outcome, and 0 being a better outcome.
Time Frame: Day 1 through Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 15 | 12 | 18 | 3
Points on a scale | 2.5 (2.3) | 3.1 (2.2) | 3.8 (3.2) | 2.7 (1.5)

9. Secondary Outcome: Duration (Hours) of Vomiting and/or Diarrhea Through Day 5
Description: The duration of diarrhea will be calculated for participants who had at least three stools classified as having loose or watery consistency, or who have at least two stools classified as having loose or watery consistency with > 300 gm of loose or watery stools in a study day (from 00:00 to 23:59). The duration will be calculated as the interval between the first time a loose/watery stool is produced on a day the participant met the criteria for diarrhea through the last loose/watery stool on a day the participant met the criteria for diarrhea. The duration of vomiting during the inpatient period will be calculated for participants who had at least two episodes of vomiting in a study day or over two consecutive days. The duration of diarrhea and/or vomiting will be calculated beginning from the first diarrheal stool or episode of vomiting until the last diarrheal stool or episode of vomiting during the inpatient period.
Time Frame: Day 1 through Day 5
Population: Modified Intention-to-Treat Population: The mITT population includes all participants who received the challenge study product and contributed both pre- and at least one post-challenge sample during the inpatient period for which a conclusion can be made regarding illness and infectivity. Participants included only experienced diarrhea and/or vomiting.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
Number analyzed (Participants) | 2 | 3 | 7 | 2
Hours
  Duration of Diarrhea: number analyzed (Participants) | 2 | 2 | 5 | 2
  Duration of Diarrhea | 11.02 (5.798) | 7.015 (4.929) | 17.264 (15.323) | 11.655 (8.733)
  Duration of Vomiting: number analyzed (Participants) | 1 | 1 | 6 | 0
  Duration of Vomiting | 2.5 (NA) — There was no standard deviation as only one participant experienced vomiting | 6.62 (NA) — There was no standard deviation as only one participant experienced vomiting | 5.845 (7.646) |
  Duration of Diarrhea and/or Vomiting | 11.37 (6.293) | 6.883 (3.492) | 15.937 (13.38) | 11.655 (8.733)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 180
Arm/Group | 3.5x10^3 Copies - Secretor Positive | 3.5x10^4 Copies - Secretor Positive | 3.5x10^5 Copies - Secretor Positive | Secretor Negative
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12 | 0/18 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/18 | 0/3
Other Adverse Events (participants affected / at risk) | 11/15 | 11/12 | 15/18 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.5x10^3 Copies - Secretor Positive (N=15) | 3.5x10^4 Copies - Secretor Positive (N=12) | 3.5x10^5 Copies - Secretor Positive (N=18) | Secretor Negative (N=3)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 7 (7) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 6 (6) | 8 (8) | 13 (14) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (3) | 3 (3) | 9 (9) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bacterial Vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Diastolic Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Diastolic Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Systolic Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Systolic Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 6 (6) | 7 (7) | 7 (7) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 7 (7) | 8 (8) | 9 (9) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 11 (11) | 0 (0)
Malaise (General disorders) | 5 (5) | 9 (9) | 9 (9) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 8 (8) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 6 (6) | 11 (11) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT04174560/Prot_001.pdf
  • Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT04174560/SAP_002.pdf
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT04174560/ICF_000.pdf